CLINICAL TRIAL: NCT02248766
Title: Clinical Performance of Habitual Wearers of Avaira Toric (Enfilcon A) When Refitted With Clariti Toric (Somofilcon A) Lenses for 1 Month.
Brief Title: Clinical Performance of Habitual Wearers of Avaira Toric When Refitted With Clariti Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-53
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- enfilcon A (Active Comparator): All participants are habitual wearers of enfilcon A lens who are refitted with somofilcon A lens
  Interventions: Device: somofilcon A
- somofilcon A (Experimental): All participants are habitual wearers of enfilcon A lens who are refitted with somofilcon A lens
  Interventions: Device: somofilcon A

INTERVENTIONS:
Device: somofilcon A — somofilcon A lens

SUMMARY:
The aim of this dispensing study is to evaluate the clinical performance of existing wearers of Avaira toric lenses following a refit with Clariti toric over 1 month of daily wear.

DETAILED DESCRIPTION:
This is a 30-subject, prospective dispensing study comparing the clinical performance of the subjects' habitual Avaira toric lenses following a refit with Clariti toric lenses. Subject's habitual Avaira toric lenses will be evaluated at the first visit and then re-fitted with a pair of Clariti toric lenses for 1 month of daily wear. After the dispensing visit, subjects will return for evaluations at 1 week, 2 weeks and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted Avaira toric contact lens (CL) wearer (at least 1 week of wear in Avaira toric)
* Has a contact lens spherical prescription between +6.00 to - 8.00 (inclusive)
* Have no less than 0.75D of astigmatism and no more than 1.75 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Is not a habitual wearer of Avaira toric lenses
* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -1.75 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, OD, Principal Investigator — Optometry Research Group (GIO)
Locations (1):
- Optometry Research Group (GIO) - Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Enfilcon A / Somofilcon A: All participants are habitual wearers of enfilcon A lens and who are refitted with somofilcon A lens
  enfilcon A: All participants wear habitual enfilcon A lens first and then refitted with somofilcon A lens
  somofilcon A: All participants wear habitual enfilcon A lens first and then refitted with somofilcon A lens
Period: Overall Study
Arm/Group | Enfilcon A / Somofilcon A
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study had a total of 30 participants. The 30 participants were evaluated with the habitual lenses (enfilcon A) and then evaluated with the (somofilcon A) lenses.
Arm/Group | Enfilcon A / Somofilcon A
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Region of Enrollment [Number; unit: participants]
  Spain | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Enfilcon A and Somofilcon A
Description: Monocular and binocular logMAR visual acuity for enfilcon A / somofilcon A assessed at baseline and somofilcon A lenses assessed at 1 week, 2 week, 4 week.
Time Frame: Baseline, 1 week, 2 week, 4 week
Measure: Mean (Standard Deviation); unit: logMar
Groups:
- Enfilcon A: All participants are habitual wearers of enfilcon A lens and who are refitted with somofilcon A lens
  enfilcon A: All participants wear habitual enfilcon A lens first and then refitted with somofilcon A lens
- Somofilcon A at 1 Week; Somofilcon A at 2 Week; Somofilcon A at 4 Week: All participants are habitual wearers of enfilcon A lenses and who are then refitted with somofilcon A lenses.
Arm/Group | Enfilcon A | Somofilcon A at 1 Week | Somofilcon A at 2 Week | Somofilcon A at 4 Week
Number analyzed (Participants) | 30 | 30 | 30 | 30
logMar
  Oculus Dexter (OD) | -0.013 (0.03) | -0.013 (0.03) | -0.010 (0.03) | -0.023 (0.03)
  Oculus Sinister (OS) | -0.010 (0.03) | -0.010 (0.03) | -0.017 (0.03) | -0.017 (0.03)
  Binocular | -0.033 (0.05) | -0.033 (0.05) | -0.040 (0.05) | -0.040 (0.05)

2. Primary Outcome: Subjective Assessments- Enfilcon A and Somofilcon A
Description: Subjective assessments for: comfort, dryness, handling, overall lens fit, and overall vision satisfaction. Enfilcon A was assessed at baseline and somofilcon A lenses assessed at 1 week, 2 week, 4 week. Scale(s): comfort (0=very poor; 10=excellent), dryness (0=very dry; 10=no dryness), handling (0=very difficult; 10=very easy), overall lens fit (0=very unstable; 10=very stable), overall vision satisfaction (0=very unsatisfied; 10=very satisfied)
Time Frame: Baseline, 1 week, 2 week, 4 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enfilcon A | Somofilcon A at 1 Week | Somofilcon A at 2 Week | Somofilcon A at 4 Week
Number analyzed (Participants) | 30 | 30 | 30 | 30
units on a scale
  Comfort on insertion | 8.53 (1.00) | 8.43 (0.62) | 8.07 (0.64) | 7.50 (0.86)
  Comfort prior to removal | 8.13 (0.94) | 7.83 (0.80) | 7.20 (0.71) | 6.70 (0.99)
  Comfort overall | 8.10 (0.92) | 7.63 (0.77) | 7.10 (0.76) | 6.20 (1.10)
  Dryness during the day | 8.47 (0.73) | 8.27 (0.64) | 7.63 (0.88) | 7.43 (1.13)
  Dryness prior to removal | 8.23 (0.73) | 8.00 (0.79) | 7.33 (0.80) | 7.03 (0.96)
  Overall dryness | 8.03 (0.67) | 7.77 (0.73) | 7.13 (0.86) | 6.70 (1.23)
  Handling | 9.23 (0.63) | 9.20 (0.55) | 9.17 (0.46) | 9.00 (0.53)
  Overall lens fit | 7.93 (0.69) | 7.90 (0.78) | 7.77 (0.76) | 8.13 (0.70)
  Overall vision satisfaction | 8.30 (0.79) | 8.10 (0.69) | 7.60 (0.67) | 7.77 (0.62)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Somofilcon A: All participants are habitual wearers of enfilcon A lens and who are refitted with somofilcon A lens
  somofilcon A: All participants wear habitual enfilcon A lens first and then refitted with somofilcon A lens
Arm/Group | Enfilcon A | Somofilcon A
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.